CLINICAL TRIAL: NCT01663675
Title: Trisomy 21 in Adulthood. Evaluation of Health and Social State in Alsace (North-eastern France)
Brief Title: Trisomy 21 in Adulthood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5249
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Down Syndrome
Keywords: Down syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Karyotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trisomy 21 (Down syndrome): Trisomy 21 (Down syndrome)
  Interventions: Genetic: karyotype

INTERVENTIONS:
Genetic: karyotype

SUMMARY:
Trisomy 21 or Down syndrome, is the most common genetic cause of cognitive disability. Currently, in Alsace, the birth prevalence is about 1 in 1600 live births, which means 10 liveborns with Down syndrome each year.If screening and prenatal diagnosis of children with trisomy 21, as well as medical care, social and educational integration in childhood was the subject of much research and has led to remarkable progress in terms of health and medical care, it is not the same for the knowledge about adolescents and adults.Despite a more and more higher life expectancy, the evolution of trisomy 21 in adulthood is often marked by a deterioration in health status, with a regression of acquired psychomotor skills, often attributed only to the precocious occurrence of Alzheimer's dementia. Nevertheless, it seems that the diagnosis of Alzheimer's dementia is often overdiagnosed, and it is well established that only a fraction of Down syndrome patients will develop this type of dementia. Too often a decline in general health, behavioral changes and decreased cognitive abilities are only attributed to the Down syndrome with an early dementia without looking for an underlying, potentially curable, disease.This study aims to better evaluate the health and social status of 100 adults with trisomy 21 in Alsace. The medical evaluation will include a comprehensive assessment of health status and quality of life conducted by the geneticist, a cardiac, sensory, hormonal, biological and radiological evaluation. A speech-language and psychomotor evaluation will also be conducted. A psychiatric consultation and a psychometric assessment will aim to assess cognitive function and to search for associated mood disorders.The expected results are to better know the natural history of trisomy 21 in adulthood, with the determination of the frequency of morbid events specific to adulthood, and also to improve the medical and paramedical care with the establishment of a monitoring program to prevent the occurrence of these morbid events.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman older than 18 years
* Down syndrome (clinical diagnosis, eventually confirmed by blood karyotype)

Exclusion Criteria:

* children
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with trisomy 21 older than 18 years living in Alsace Region (North-eastern France)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ALEMBIK Yves, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Dieudonne Y, Uring-Lambert B, Jeljeli MM, Gies V, Alembik Y, Korganow AS, Guffroy A. Immune Defect in Adults With Down Syndrome: Insights Into a Complex Issue. Front Immunol. 2020 May 8;11:840. doi: 10.3389/fimmu.2020.00840. eCollection 2020. PMID 32457756
- [Derived] Guffroy A, Dieudonne Y, Uring-Lambert B, Goetz J, Alembik Y, Korganow AS. Infection risk among adults with down syndrome: a two group series of 101 patients in a tertiary center. Orphanet J Rare Dis. 2019 Jan 11;14(1):15. doi: 10.1186/s13023-018-0989-x. PMID 30634988